CLINICAL TRIAL: NCT06570824
Title: Network Based Repetitive Transcranial Magnetic Stimulation (rTMS) as an Intervention for Levodopa-induced Dyskinesia (LID) in Parkinson's Disease (PD)
Brief Title: rTMS as an Intervention for Levodopa-induced Dyskinesia
Acronym: ADAPT-LIDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Responsible Party: Principal Investigator, Hartwig R. Siebner, Head of Research, Prof, DMSc, Danish Research Centre for Magnetic Resonance
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ADAPT-LIDI
Record Dates: First submitted 2024-05-03; First posted 2024-08-26 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Dyskinesia, Drug-Induced; Parkinson Disease
Keywords: Basal Ganglia Diseases; Parkinson's Disease; Central Nervous System Diseases; Movement Disorders; Synucleinopathies; Neurodegenerative Diseases; Dyskinesias; LID; Levodopa induced dyskinesia; Pre-SMA
MeSH Terms: conditions — Dyskinesia, Drug-Induced; Parkinson Disease; Basal Ganglia Diseases; Central Nervous System Diseases; Movement Disorders; Synucleinopathies; Neurodegenerative Diseases; Dyskinesias

STUDY DESIGN:
Intervention Model Description: The study has a double-blinded crossover design. The research participants will, in two separate stimulation sessions, receive either real rTMS treatment or a sham-TMS stimulation. The session order (real rTMS first or sham first) will be randomised between research participants. The research participant will be blinded to which treatment (real or sham) they receive at any session. There will be two sequential groups of patients. First group will receive gamma burst rTMS stimulation and sham and the other group will receive beta burst rTMS and sham.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will receive sham rTMS by flipping the coil upside down. This will still provide similar sensory experience as an active stimulation that the patients will not distinguish between. Dyskinesia assessment is filmed during the visit and an experienced rater is unaware of a treatment condition of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gamma burst rTMS (Active Comparator): Real stimulation with 4 pulses at the frequency of 130Hz repeating at 1 Hz will be delivered on the pre-SMA using the active side of the coil for 30 minutes
  Interventions: Device: active TMS
- Sham gamma burts rTMS (Sham Comparator): Sham stimulation with 4 pulses at the frequency of 130Hz repeating at 1Hz will be delivered on the pre-SMA with a non-active side of the coil for 30 minutes
  Interventions: Device: sham TMS
- Beta burst rTMS (Active Comparator): Real stimulation with 4 pulses at the frequency of 20Hz repeating at 1 Hz be delivered on the pre-SMA using the active side of the coil for 30 minutes
  Interventions: Device: active TMS
- Sham beta burst rTMS (Sham Comparator): Sham stimulation with 4 pulses at the frequency of 20Hz repeating at 1Hz will be delivered on the pre-SMA with a non-active side of the coil for 30 minutes
  Interventions: Device: sham TMS

INTERVENTIONS:
Device: active TMS — Transcranial magnetic stimulation using MagVenture XP Orange Stimulator using active side of MagVenture Cool-B70 coil
  Arms: Beta burst rTMS; Gamma burst rTMS
Device: sham TMS — Sham transcranial magnetic stimulation using MagVenture XP Orange Stimulator, flipping the active side of the MagVenture Cool-B70 coil
  Arms: Sham beta burst rTMS; Sham gamma burts rTMS

SUMMARY:
The proposed study investigates the use of repetitive transcranial magnetic stimulation (rTMS) as a treatment for levodopa-induced dyskinesia (LID) in Parkinson's Disease (PD). Specifically, the study aims to determine whether patterned stimulation of the pre-supplementary motor area (pre-SMA) can delay the onset of LID after levodopa intake and reduce LID severity in PD patients. This study will provide critical insights into potential targets for rTMS treatment, optimal rTMS parameters, and the mechanisms underlying LID in Parkinson's disease.

DETAILED DESCRIPTION:
Long-term use of levodopa in Parkinson's Disease (PD) often leads to motor complications, such as Levodopa-Induced Dyskinesia, which significantly impacts patients' daily lives. Various brain regions have been targeted for treatment with Transcranial Magnetic Stimulation (TMS), including the supplementary motor area (SMA), primary motor cortex, cerebellum, and prefrontal cortex. Specifically, targeting the pre-SMA with 1-Hz rTMS has been shown to delay and reduce dyskinesia severity in PD patients following levodopa administration. These findings suggest that the pre-supplementary motor area is a promising target for brain stimulation therapy, as it plays a causal role in the pathophysiology of peak-of-dose dyskinesia.

The current study aims to build on previous research by optimizing the stimulation intensity and location based on individual neuroanatomy and simulated electric fields. Additionally, the study will explore the impact of rTMS delivered in short high-frequency bursts, differing from the single rTMS pulses used in previous studies. In the context of LID, Deep Brain Stimulation (DBS) typically targets the subthalamic nucleus (STN) using gamma frequencies (40-200 Hz, most commonly 130 Hz). Drawing from this principle, the study posits that delivering rTMS bursts at gamma frequencies to the pre-SMA will effectively mitigate LID symptoms. Moreover, evidence from cortical brain rhythm recordings highlights that beta frequencies (12-30 Hz), which are crucial for movement control and are disrupted in PD, may also hold therapeutic potential. Therefore, the study will investigate whether rTMS bursts at beta frequencies could similarly reduce LID symptoms. Given the absence of prior research directly comparing the effects of different burst frequencies on LID, the study will systematically apply two distinct burst frequencies, in separate patient groups, to determine which, if either, produces a meaningful reduction in LID symptoms.

Dyskinesia onset time and severity will be measured using the Unified Dyskinesia Rating Scale (UDysRS) and assessed by a clinician rater who is blinded to the treatment condition. The results will be compared between the active and sham stimulation conditions.

ELIGIBILITY:
Inclusion Criteria:

* Clinically established or probable PD
* Clinical Diagnostic Criteria for Parkinson's Disease
* Peak-of-dose levodopa-induced dyskinesia.
* Stable antiparkinsonian medicine for at least four weeks.
* Signed informed consent.

Exclusion Criteria:

* Psychiatric disorders.
* Usage of antipsychotic medication, Donepezil, and GABAergic medications (such as pregabalin and gabapentin).
* Regular usage of benzodiazepines and opioids (more than once per week).
* History of neurological disease other than Parkinson's disease.
* History of epilepsy/conditions associated with increased risk to seizure-induction through TMS.
* Close relatives suffering from epilepsy/conditions associated with increased risk to seizure-induction through TMS.
* Contraindications for MRI scan
* Female participants of childbearing age must not be pregnant and that they must use contraception during the trial.
* Refuse to be informed about new health related information and accidental health related findings that might appear through participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Unified Dyskinesia Rating Scale (UDysRS) | Baseline (usual medication intake) and up to 40 minutes after taking 150 % of normal morning levodopa dose as Madopar Quick
  UDysRS utilizes rater information, patient self-report and objective measures of dyskinesia to provide assessments of impairment and disability due to dyskinesia.The UDysRS total score ranges from 0 to 104 with a lower score indicating less dyskinesia.
Dyskinesia onset time | Baseline (usual medication intake) and up to 40 minutes after taking 150 % of normal morning levodopa dose as Madopar Quick
  The onset time of dyskinesia in minutes after levodopa administration

SECONDARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline (usual medication intake) and up to 40 minutes after taking 150 % of normal morning levodopa dose as Madopar Quick
  Measure the changes of scores of United Parkinson's Disease Rating Scale Part III in active stimulation compared to sham. The total scores range from 0 (good health) to 132 (poor health).

OTHER OUTCOMES:
TMS adverse events and associated sensations questionnaire (TMSens_Q) | Immediately after the TMS intervention (sham and active)
  Questionnaire for assessing any side effects and sensations associated with TMS stimulation, including the assessment of masking (sham or active treatment) of participants.
Transcranial evoked potentials (TEPs) | Before and immediately after the TMS intervention (sham and active), up to 20 minutes after taking 150 % of normal morning levodopa dose as Madopar Quick
  Change in cortical excitability pre-post stimulation and OFF-ON states after levodopa administration
Event related potentials (ERPs) | Immediately after taking 150 % of normal morning levodopa dose as Madopar Quick
  Dynamics of EEG during a Go/Nogo task: movement related potentials, spectral features
Non-Motor Symptoms Scale for Parkinson's Disease (NMSS) | Baseline, 4-8 weeks after inclusion
  The Non-Motor Symptoms Scale (NMSS) is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The scores on the NMSS range from 0 to 360, with higher scores implying a higher severity and frequency of nonmotor symptoms.
Non-Motor Fluctuation Assessment (NoMoFA) Questionnaire | Baseline, 4-8 weeks after inclusion
  27-item self-administered questionnaire that is used for capturing both static and fluctuating non-motor symptoms in PD. Possible score for the NoMoFA ranges from 0 to 81 points, with higher scores implying a higher severity and frequency of nonmotor symptoms.
CANTAB battery | Baseline, 4-8 weeks after inclusion
  Measures of response inhibition, spatial planning and working memory and reaction time
The Parkinson's Disease Questionnaire (PDQ-39) | Baseline, 4-8 weeks after inclusion
  39 item self-administered questionnaire that assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better quality of life.
The World Health Organization Quality of Life (WHOQOL) | Baseline, 4-8 weeks after inclusion
  General quality of life assessment as a part of patient reported outcome assessment. The possible score ranges in each case from 0 to 100 points. Higher scores indicate better quality of life.
Movement dynamics | Continuous up to 8 weeks after inclusion
  Duration of dyskinesia per day in minutes, OFF/ON periods per day in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig R. Siebner, Prof., Principal Investigator — Head of Research, Prof, DMSc
Locations (1):
- DRCMR, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Sharing of anonymised data
Time Frame: After study completion
Access Criteria: Anonymised data, reasonable request

REFERENCES:
- [Background] Lohse A, Meder D, Nielsen S, Lund AE, Herz DM, Lokkegaard A, Siebner HR. Low-frequency transcranial stimulation of pre-supplementary motor area alleviates levodopa-induced dyskinesia in Parkinson's disease: a randomized cross-over trial. Brain Commun. 2020 Sep 18;2(2):fcaa147. doi: 10.1093/braincomms/fcaa147. eCollection 2020. PMID 33225277
- [Background] Herz DM, Haagensen BN, Christensen MS, Madsen KH, Rowe JB, Lokkegaard A, Siebner HR. The acute brain response to levodopa heralds dyskinesias in Parkinson disease. Ann Neurol. 2014 Jun;75(6):829-36. doi: 10.1002/ana.24138. Epub 2014 May 28. PMID 24889498
- See also: Institutional website — http://drcmr.dk